CLINICAL TRIAL: NCT00817648
Title: A 6-Week, Multicenter, Rater-blind, Randomized, Risperidone-controlled Study to Evaluate the Efficacy and Safety of Seroquel (Quetiapine Fumarate) in the Treatment of Chinese Han Patients With Schizophrenia
Brief Title: A Study to Evaluate the Efficacy and Safety of Seroquel in Chinese Han Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: LI, Huafang, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1443L00071; SMHC-098
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Schizophrenia
Keywords: schizophrenia; antipsychotics; quetiapine; risperidone; efficacy; safety; multicenter; rater-blind; randomized; chinese; han
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate; Risperidone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Quetiapine fumarate, flexible doses(600-750 mg/d)
  Interventions: Drug: Quetiapine
- 2 (Active Comparator): risperidone, flexible doses(3-6 mg/d)
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: Quetiapine — Quetiapine fumarate, 25mg/200 mg, the dose titration is carried in week 1. flexible doses(600-750 mg/d) from week 2 to week 6. If a patient is intolerant, the doses can be adjusted as judged by investigator.
  Other Names: Seroquel
  Arms: 1
Drug: risperidone — risperidone, 1mg/tablet, the dose titration is carried in week 1. flexible doses(3-6 mg/d) from week 2 to week 6. If a patient is intolerant, the doses can be adjusted as judged by investigator.
  Other Names: Risperdal
  Arms: 2

SUMMARY:
The primary objective of this study is to evaluate the efficacy of seroquel in the treatment of patients with acute schizophrenia compared with risperidone by evaluating the change of PANSS total score from the baseline to week 6.

DETAILED DESCRIPTION:
This is a rater- blind, parallel assignment, randomized and active controlled study. The subjects investigated are outpatients or inpatient with schizophrenia from the Chinese Han race. The screening phase lasts for 1 week. The eligible patients enter the next randomized treatment phase. The titration duration is 1 week. After the first week, the patients are administered with a flexible dose regimen. In this study, the effective doses range of seroquel and risperidone are 600-750mg/d and 3-6mg/d respectively and the treatment duration lasts for 6 weeks.

The efficacy and safety of seroquel in the treatment of patients with schizophrenia have been confirmed by multiple double blind studies. This study is designed to evaluate the efficacy and safety of seroquel in the treatment of Chinese Han patients with schizophrenia. Therefore, the single blind and active control design should be selected for this study. The drug titration method and dose are within the range specified in the instruction and patients with schizophrenia are tolerant to the drug in clinical treatment.

The purpose of schizophrenic patient treatment is to improve the core symptoms, prevent suicide and other aggressive behavior, alleviate the side reactions caused by the drug, and recover the life functions of patients. Generally, the treatment in the acute phase lasts for 6 to 8 weeks. In this study, the treatment in the acute phase lasts for 6 weeks.

The rating scales used in this study are standard psychiatric rating scales with good validity and are widely used in the study of antischizophrenia drugs and in the treatment of patients with schizophrenia in China. The PANSS is developed from two early rating scales, namely the brief psychiatric rating scale (BPRS) and the psychiatric rating scale. The high inter-investigator reliability and repeated measurement reliability of these scales have been proved by multiple studies. The clinical global impression (CGI) is a simple but convenient global impression scale. It is applicable to any patients treated and studied by the psychiatric department. The Carlgary depression scale for schizophrenia (CDSS) is used to evaluate the depressive symptoms of patients with schizophrenia. It has good reliability and validity. The abnormal involuntary movement scale (AIMS) is another evaluation tool consisting of 12 items. The AIMS is used to evaluate the abnormal involuntary movements related to antischizophrenia drugs. The AIMS is nearly the most frequently used multi-item rating scale evaluating of tardive dyskinesia. The Simpson and Angus scale (SAS) is also a rating scale commonly used since its release in 1970. The validity of SAS has been verified in the double blind and placebo-controlled study involving two haloperidol doses.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent provided by legal guardians or patients.
2. Patients who met DSM-IV criteria for schizophrenia: 295.20 (Schizophrenia, Catatonic Type), 295.10 (Schizophrenia, Disorganized Type), 295.30 (Schizophrenia, Paranoid Type), 295.60 (Schizophrenia, Residual Type), and 296.90 (Mood Disorder NOS).
3. Age from 18-65 years old, male or female, Han nationality.
4. PANSS total score at least 70 at baseline.
5. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment.
6. Able to understand and comply with the requirements of the study. -

Exclusion Criteria:

1. Pregnancy or lactation.
2. A diagnosis of any DSM-IV Axis I disorders that is not defined in the inclusion criteria, except schizophrenia.
3. Patients who have an imminent risk of suicide or a danger to self or others as judged by investigator.
4. Known intolerance or lack of efficacy to seroquel and/or risperidone, as judged by the investigator.
5. Use of seroquel and/or risperidone within 28 days prior to enrolment.
6. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir.
7. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids.
8. Use of a long acting antipsychotics Within one dosing interval
9. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria.
10. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse as defined by DSM-IV criteria within 28 days prior to enrolment.
11. Medical conditions that would affect the absorption, distribution, metabolism, or excretion of study treatment.
12. Unstable or inadequately treated medical illness (e.g. CHF - congestive heart failure, angina pectoris, hypertension) as judged by the investigator.
13. Involvement in the planning and conduct of the study.
14. Participation in another drug trial within 28 days prior enrolment into this study.
15. Patient with diabetes mellitus.
16. The patient's absolute neutrophil count (ANC) ≤ 1.5 x 109/L and the ALT and AST values in the liver function test exceeding two times of the upper limits of normal values.
17. Use of Electroconvulsive therapy within 28 days prior to randomization.
18. Use of clozapine within 28 days prior to randomization.
19. Previous enrolment in the present study -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
the change of PANSS total score | from the baseline to week 6

SECONDARY OUTCOMES:
The Carlgary depression scale for schizophrenia (CDSS) | from the baseline to week 6
The abnormal involuntary movement scale (AIMS) | from the baseline to Week 6
The Simpson and Angus scale (SAS) | from the baseline to week 6
The clinical global impression (CGI),including CGI-I and CGI-S | from the baseline to week 6

CONTACTS AND LOCATIONS:
Overall Officials: Huafang LI, MD,PhD, Principal Investigator — Drug Clinical Trial Office, Shanghai Mental Health Center
Locations (4):
- China (4):
  - Mental Health Center of Luwan District, Shanghai, Shanghai Municipality
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Branch Hospital of Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Huzhou Third People Hospital, Huzhou, Zhejiang

REFERENCES:
- [Background] Mandrioli R, Fanali S, Ferranti A, Raggi MA. HPLC analysis of the novel antipsychotic drug quetiapine in human plasma. J Pharm Biomed Anal. 2002 Nov 7;30(4):969-77. doi: 10.1016/s0731-7085(02)00395-3. PMID 12408887
- [Background] Davis PC, Wong J, Gefvert O. Analysis and pharmacokinetics of quetiapine and two metabolites in human plasma using reversed-phase HPLC with ultraviolet and electrochemical detection. J Pharm Biomed Anal. 1999 Jun;20(1-2):271-82. doi: 10.1016/s0731-7085(99)00036-9. PMID 10704032
- [Background] Riedel M, Muller N, Strassnig M, Spellmann I, Engel RR, Musil R, Dehning S, Douhet A, Schwarz MJ, Moller HJ. Quetiapine has equivalent efficacy and superior tolerability to risperidone in the treatment of schizophrenia with predominantly negative symptoms. Eur Arch Psychiatry Clin Neurosci. 2005 Dec;255(6):432-7. doi: 10.1007/s00406-005-0622-6. Epub 2005 Nov 4. PMID 16267634
- [Background] Buckley PF. Efficacy of quetiapine for the treatment of schizophrenia: a combined analysis of three placebo-controlled trials. Curr Med Res Opin. 2004 Sep;20(9):1357-63. doi: 10.1185/030079904125004510. PMID 15383183
- [Result] Miodownik C, Lerner V. Quetiapine: efficacy, tolerability and safety in schizophrenia. Expert Rev Neurother. 2006 Jul;6(7):983-92. doi: 10.1586/14737175.6.7.983. PMID 16831113